CLINICAL TRIAL: NCT06363929
Title: A Study to Evaluate the Accuracy of Continuous Glucose Monitors in Neonates With Hyperinsulinism.
Brief Title: Continuous Glucose Monitoring in Neonatal Hyperinsulinism
Status: Terminated | Type: Observational
Why Stopped: Principal investigator is leaving the study.
Sponsor: MemorialCare Health System (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 341-23
Record Dates: First submitted 2023-12-20; First posted 2024-04-12 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hyperinsulinism; Hypoglycemia Neonatal
MeSH Terms: conditions — Hyperinsulinism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Neonates with hyperinsulinism: Neonates with a diagnosis of hyperinsulinism will wear a Dexcom G6 continuous glucose monitor placed for 10 days.
  Interventions: Device: Dexcom G6 continuous glucose monitor

INTERVENTIONS:
Device: Dexcom G6 continuous glucose monitor — Dexcom G6 continuous glucose monitor to be placed on neonates with hyperinsulinism for 10 days.

SUMMARY:
The investigators are studying the accuracy of Dexcom G6 continuous glucose monitors placed on babies with hyperinsulinism in the Miller Children's Hospital Neonatal Intensive Care Unit. The participants will wear the device for 10 days on their lateral thigh. Whenever blood sugars are checked by glucometer, the investigators will also record the continuous glucose monitor sugar. Additionally, if the continuous glucose monitor alarms for a low sugar or an impending low sugar, the investigators will check the blood sugar by glucometer and, if verified to be low, treat the low blood sugar accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Age: 0-90 days old
* Gestational Age: > 28 weeks gestational age
* Diagnosis of hyperinsulinism based on critical sample and/or glucagon challenge

Exclusion Criteria:

* Diffuse skin disease such that placement of a Dexcom G6 sensor would be difficult to secure
* Infants colonized or infected with multi-drug resistant organisms (i.e. MRSA, VRE, ESBL producing bacteria)
* Infants on hypothermic protocols
* Infants expected to remain in the NICU <24 hours
* Infants enrolled in a competing clinical trial
* Family/team have decided to limit or redirect from aggressive NICU technological support
* Ward of the state

Ages: 24 Hours to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates with hyperinsulinism in the Miller Children's Hospital Neonatal Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Mean absolute relative difference (MARD) | Through study completion, about 2 years
  Mean absolute relative difference (MARD) between Dexcom G6 glucoses and point of care blood or plasma glucoses.

SECONDARY OUTCOMES:
Mean absolute difference (MAD) | Through study completion, about 2 years
  MAD between Dexcom G6 glucoses and the point of care blood or plasma glucoses and the percentage of Dexcom G6 glucose values within 15 mg/dL, 20 mg/dL and 30 mg/dL of point of care blood or plasma glucose values when they are <100 mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Erin L Okawa, MD, Principal Investigator — Memorial Health Services
Locations (1):
- Miller Children's Hospital, Long Beach, California, United States